CLINICAL TRIAL: NCT00860080
Title: A First in Man, Phase I, Single-blind, Placebo-controlled Study Investigating the Local Tolerability, Safety and Pharmacokinetics in Three Doses of PXL01 and Placebo in 15 Healthy Volunteers
Brief Title: Safety Study Investigating Local Tolerability and Pharmacokinetics of PXL01 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaSurgics AB (Industry)
Responsible Party: Margit Mahlapuu/CSO, PharmaSurgics AB
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PHSU01; EudraCT number: 2008-007506-11
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Post-surgery Adhesion Formation
Keywords: post-surgery adhesion formation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PXL01 (Experimental): Four Subjects per cohort will receive 10, 20, or 40 mg PXL01 respectively.
  Interventions: Drug: PXL01
- Placebo (Placebo Comparator): One subject per cohort will receive 10, 20, or 40 mg Placebo respectively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PXL01 — PXL01 is a synthetic peptide sequentially derived from human lactoferrin. The substance is formulated in a viscous solution of sodium hyaluronate. 10, 20, and 40 mg PXL01 will be administered as an abdominal subcutaneous injection of 0.5, 1, and 2 ml respectively.
  Arms: PXL01
Drug: Placebo — Placebo is prepared by dilution of sodium hyaluronate using 0.9% sodium chloride solution. The concentration of sodium hyaluronate is 15 mg/ml after dilution. Placebo will be administered as an abdominal subcutaneous injection of 0.5, 1, and 2 ml respectively.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine whether three different single doses of PXL01 are safe and well tolerated by healthy volunteers. The pharmacokinetic properties of PXL01 (same doses) will also be investigated.

DETAILED DESCRIPTION:
The primary objective is to investigate the local tolerability and safety of PXL01 in the doses 10, 20, 40 mg, and placebo. The secondary objective is to investigate the pharmacokinetic properties of PXL01 in single doses of 10, 20, and 40 mg.

This is a single-blind, placebo-controlled, single dose administration study in male healthy volunteers. Each Subject will visit the centre three times; one screening visit, one dose administration visit and one follow-up visit over a period of approximately 3 weeks.

At Visit 1 (screening visit), the Subject will be given verbal and written patient information and the informed consent will be signed. Thereafter, the Subject will be assessed for eligibility. Demography, concomitant medication, and medical history will be documented. A physical examination will be performed and blood/urine will be collected for safety analysis. Tests for HIV, Hepatitis B and C, drug screening and alcohol breath test will be performed. Vital signs and a 12-lead ECG will be recorded.

At Visit 2 (dose administration visit), which will occur 7±3 days after the screening visit, the Subjects will first perform an alcohol breath test and PXL01/placebo will then be administered as an abdominal subcutaneous injection. Blood samples for pharmacokinetic analysis will be drawn, pulse and blood pressure will be recorded, and local tolerability assessments will be performed prior to and 15min, 30min, 45min, 60min, 1h 15min, 1h 30min, 2h, 4h, 8h and 24h after the injection. A 12-lead ECG and body temperature will be recorded prior to dose, 1h, 2h, 4h, 8h and 24h after the injection. Blood will be collected prior to and 24 hours after the injection. Adverse Events (AEs) will be recorded and telemetry heart rythm will be monitored continuously. The Subjects will stay at the clinic for about 26 hours after the injection.

Visit 3 (Follow-up visit) will be performed 5-8 days after Visit 2. A physical examination and local tolerability assessments will be performed. Vital signs, a 12-lead ECG and AEs will be recorded. Blood/urine will be collected for safety analysis.

Each group will start by dosing two Subjects. One Subject will receive placebo and the other active treatment. If there are no safety/tolerability concerns within 48 hours, another three Subjects will receive the dose.

Prior to dose escalation, a safety monitoring board will discuss all safety data. In case of any safety/tolerability concerns, dosing may be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Male healthy volunteers
2. Age ≥ 18 to ≤ 50 years
3. BMI ≥ 18.5 to ≤ 30.0 kg/m2
4. Signed written informed consent
5. Ability to co-operate

Exclusion Criteria:

1. Concomitant treatment with any drug within 7 days of dosing. This includes prescription and OTC drugs, as well as herbal medicines. Exceptions are occasional intake of paracetamol (maximum 1,500 mg/day; and not exceeding 3,000 mg/week) and nasal sprays, at the discretion of the Investigator
2. Known allergy or hypersensitivity to PXL01, sodium hyaluronate, or structurally related compounds
3. Known allergies to avian proteins, feathers, and egg products
4. Enrolment in any other clinical study within 3 months prior to screening visit, or previous participation in the present study
5. Drug and/or alcohol abuse
6. Use of any nicotine containing products within one month prior to the screening visit
7. Scar tissue at the planned injection site
8. History of severe drug allergy or hypersensitivity as judged by the Investigator
9. Any planned major surgery within the duration of the study
10. Any other condition or symptoms preventing the Subject from entering the study, according to the Investigator's judgement
11. Donation of blood within 3 months prior to screening
12. Positive serology for HIV, hepatitis B, and/or hepatitis C viruses
13. Positive results on drug screening

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety (the frequency and severity of adverse events, vital signs, haematology, clinical chemistry, urinalysis, electrocardiogram) and local tolerability (inspection of the injection site) | From dosing until 2 weeks after dosing

SECONDARY OUTCOMES:
The pharmacokinetic parameters Cmax, tmax, AUC, and t1/2 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Huss, PhD, Principal Investigator — Berzelius Clinical Research Center
Locations (1):
- Berzelius Clinical Research Center, Linköping, Sweden